CLINICAL TRIAL: NCT01789866
Title: Dynamic Roles of Dietary Docosahexaenoic Acid (DHA) and Lutein in Brain Function in Healthy Children
Brief Title: DHA & Lutein and fMRI Brain Mapping in Healthy Children
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Yvonne Lamers, Principle Investigator, University of British Columbia
Other Study IDs: H12-01306
Record Dates: First submitted 2012-12-20; First posted 2013-02-12 (Estimated); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Healthy Nutrition
Keywords: DHA; lutein; neurodevelopment; fMRI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Studies suggest that lutein and n-3 fatty acids may influence the development of a child's brain and may be related to how well children learn. Both lutein and the n-3 fats (also known as omega-3 fats) are not made by the body and must be obtained in the diet. The investigators are interested to understand the importance of n-3 fats and lutein to child brain development. Functional magnetic resonance imaging (fMRI) will make it possible to look into the brain from the outside and see which parts of the brain are being used as children complete working memory tasks. The investigators will study brain function using fMRI among children with different intakes of n-3 fats and lutein.

Hypothesis:

1. Children 6 years of age consuming < 25 mg/day DHA and < 400 μg lutein/day will show poorer activation of brain areas on fMRI than children consuming > 150 mg/day DHA and > 1,200 μg/day lutein.
2. Children consuming < 400 μg lutein/day and > 150 mg/day DHA will also show differences in fMRI results when compared to children consuming > 150 mg/day DHA and > 1,200 μg/day lutein.

DETAILED DESCRIPTION:
Study Design:

A cross-sectional observational study of 62 school-age children in Vancouver, Canada.

Dietary intake assessment:

Children's dietary intake over the previous four weeks was estimated by interview with a parent using a Food Frequency Questionnaire. Three 24h recalls were administered, using the five-pass review technique. The children's dietary intake of DHA was quantified using nutrient analysis software (ESHA Food Processor SQL, version 10.10.0.0; ESHA Research), using Canadian foods, and checking the fatty acid composition of all foods and beverages for accuracy, modifying if necessary based on labels or laboratory analysis of the product.

Blood Markers EDTA venous blood was collected and was centrifuged to collect Red Blood Cells (RBC). RBC fatty acids were extracted and quantified by routine gas liquid chromatography. RBC-DHA to DPA (n-6) ratio was used as an indicator of DHA status.

Cognitive Measures The Kaufman Assessment Battery for Children (KABC)-II (Kaufman, 2004) was administered by one of two individuals trained in child psychometric testing. The KABC consists of several scales: (1) the Sequential Processing Scale measures short-term memory; (2) the Learning Ability Scale measures long-term storage and retrieval; & (3) the Simultaneous Processing Scale measures visual processing. Results of these 3 scales may be combined to give a composite Mental Performance Index (MPI) score. The Delayed Recall subtest was used to evaluate long-term memory.

Statistical Analysis DHA intake and RBC-DHA:DPA were log transformed; transformed data were used in the subsequent analyses. Pearson's correlation tests were conducted to test (1) the associations between DHA intake and RBC-DHA:DPA ratio and (2) the associations between DHA intake and RBC-DHA:DPA with KABC-II domain scores.

ELIGIBILITY:
Inclusion Criteria:

* full-term
* single birth (no multiple births)
* no major illness or surgery requiring hospitalization likely to impact the outcomes
* no metabolic, congenital or allergic disease that impact food intakes
* parents have sufficient command of English language to complete the informed consent and study documents

The specific inclusion enrollment criteria for:

Group 1: children consuming <25 mg/day DHA and < 400 μg/day lutein, n=24; Group 2: children consuming >150 mg/day DHA and >1,200 μg/day lutein, n=24; Group 3: children consuming >150 mg/day DHA and <400 μg/day lutein, n=10;

Exclusion Criteria:

* children of mothers enrolled in studies by our group that involved randomization to supplemental DHA during pregnancy
* children for whom blood, diet records or developmental tests at 5 years and 9 months of age are incomplete
* children consuming 25-150 mg/day DHA or 400-1200 μg/day lutein
* children of mothers who do not sign the informed consent
* any children having a cardiac pacemaker, aneurysm clip, cochlear implant of possible metallic foreign bodies in the eyes or other contraindication as detailed in the C&W MRI Patient Screening Form will be excluded from this study.

Ages: 69 Months to 78 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: school-age children differentiated by intake of DHA and lutein
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2012-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
fMRI data | 5 years 8 months to 6 years
  fMRI data will be collected for subjects differentiated by DHA and lutein status completing tasks for working memory, working language, visual working memory and visual acuity

SECONDARY OUTCOMES:
cognitive development with standardized developmental tests | 5 years 8 months to 6 years
  Assessment with the Kaufman Developmental Assessment Battery

OTHER OUTCOMES:
plasma lutein and Red blood cell DHA | 5 years 8 months to 6 years
  plasma lutein and red blood cell DHA biochemistries

CONTACTS AND LOCATIONS:
Overall Officials: Sheila M Innis, PhD, Principal Investigator — Child & Family Research Institute, University of British Columbia
Locations (1):
- Child & Family Resaerch Center, Vancouver, British Columbia, Canada